CLINICAL TRIAL: NCT01122433
Title: Evaluation of the C-MAC Video Laryngoscope After Failed Direct Laryngoscopy
Brief Title: Airway Management Study to Evaluate the C-MAC Video Laryngoscope as an Alternative to the Direct Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Department of Anaesthesiology, Prof. C. Werner, Universitätsmedizin of the JG University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PN-201005
Record Dates: First submitted 2010-05-05; First posted 2010-05-13 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Unexpected Difficult Airway
Keywords: difficult airway; indirect laryngoscopy; C-MAC video laryngoscope

ARMS (1):
- C-MAC (Experimental): After a maximum of three failed intubation attempts using direct laryngoscope the C-MAC video laryngoscope is used as an emergency airway device.
  Interventions: Device: Endotracheal intubation using the C-MAC video laryngoscope

INTERVENTIONS:
Device: Endotracheal intubation using the C-MAC video laryngoscope — Using the C-MAC video laryngoscope for endotracheal intubation after failed direct laryngoscopy

SUMMARY:
The purpose of this study is to evaluate the C-MAC video laryngoscope in difficult airway situations.

DETAILED DESCRIPTION:
Unanticipated difficulties during tracheal intubation and failure to intubate are among the leading causes of anaesthesia related morbidity and mortality. Using the technique of video laryngoscopy, the alignment of the oral and pharyngeal axis to facilitate endotracheal intubation is obsolete. In this study we evaluate the C-MAC video laryngoscope (STORZ, Tuttlingen, Germany) for endotracheal intubation in difficult intubation situations (Cormack & Lehane (CL) grade 3 and 4) validated by Macintosh laryngoscope. We hypothesize that endotracheal intubation is possible using the C-MAC in patients after failed direct laryngoscopy. We also examine whether visualisation of the glottis is improved with this device compared to direct laryngoscopy and possible complications such as soft tissue injury.

ELIGIBILITY:
Inclusion Criteria:

* Unexpected difficult airway

Exclusion Criteria:

* History of difficult or impossible mask ventilation
* Age < 18 years
* ASA grade > 3
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Success rate of endotracheal intubation using the C-MAC video laryngoscope
  The investigators evaluate the C-MAC as an alternative after failed direct laryngoscopy. Primary outcome measure is the success rate using the C-MAC video laryngoscope in unexpected difficult airways.

SECONDARY OUTCOMES:
- improved glottic view
  According to the Cormacl-Lehane classification the improved glottis view using the C-MAC is documented.
- complications
  Possible complications are supra glottic trauma, tooth damage, soft tissure bleeding,...
- numbers of intubation attempts
  Necessary intubation attempts using the C-MAC video laryngoscope to secutre the airway.
- size of blade (C-MAC)
  Different blades are available for the C-MAC. We evaluate with which blade securing the airway was possible.

CONTACTS AND LOCATIONS:
Overall Officials: Tim Piepho, MD, Principal Investigator — Department of Anaesthesiology, Universitätsmedizin Mainz; Rüdiger R Noppens, MD, Principal Investigator — Department of Anaesthesiology, Universitätsmedizin Mainz
Locations (1):
- Univeritätsmedizin of the JG University, Department of Anaesthesiology, Mainz, Germany